CLINICAL TRIAL: NCT00799942
Title: Long-term Open-label Extension Study to Assess the Safety, Tolerability, and Efficacy of Neramexane Mesylate in Congenital Idiopathic Nystagmus and Acquired Nystagmus
Brief Title: Open-lable Extension Study on Safety and Efficacy of Neramexane to Treat Congenital and Acquired Nystagmus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 92579-0738/1; 2007-007663-25
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Nystagmus, Congenital; Nystagmus, Acquired; Multiple Sclerosis
Keywords: Nystagmus, congenital idiopathic
MeSH Terms: conditions — Nystagmus, Congenital; Nystagmus, Pathologic; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Neramexane mesylate — open-label treatment of 36 months Neramexane mesylate up to 75 mg per day

SUMMARY:
The purpose of this study is to investigate the long-term safety, tolerability and efficacy of neramexane mesylate in the treatment of congenital idiopathic nystagmus (CIN). In addition, a subgroup of multiple sclerosis (MS) patients suffering from acquired nystagmus will be included.

ELIGIBILITY:
Inclusion Criteria:

* patients who has succesfully completed the lead-in study MRZ 92579-0707/1

Exclusion Criteria:

* Occurence of any major treatment-emergent adverse event or condition during the previous protocol (MRZ 92579-0707/1)

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
Long-term safety, Visual acuity | Baseline, week 4, month 3, 6, 9, 12, 18, 24, 30, 36 and follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester Royal Infirmary, Ophthalmology Group, Leicester, United Kingdom